CLINICAL TRIAL: NCT05622149
Title: Is Strength Training a Viable Exercise Modality for Fat Loss?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: City University of New York (Other)
Responsible Party: Principal Investigator, Todd Miller, Prinicipal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011638
Record Dates: First submitted 2018-03-19; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
Keywords: resistance training; metabolism
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention
- Diet Only (Experimental): Subjects were given calorie and macronutrient intake goals and were told to hit those goals as closely as possible on a daily basis for 16 weeks.
  Interventions: Behavioral: Diet Only
- Training Only (Experimental): Subjects were given a 3 times per week supervised resistance training program for 16 weeks
  Interventions: Behavioral: Training Only
- Diet plus Training (Experimental): Subjects were given calorie and macronutrient intake goals and were told to hit those goals as closely as possible on a daily basis for 16 weeks. Subjects were given a 3 times per week supervised resistance training program for 16 weeks
  Interventions: Behavioral: Diet plus Training

INTERVENTIONS:
Behavioral: Diet Only — Food tracking based on macronutrient goals.
  Arms: Diet Only
Behavioral: Training Only — Subjects completed 16 weeks of supervised resistance training
  Arms: Training Only
Behavioral: Diet plus Training — Food tracking plus resistance training.
  Arms: Diet plus Training

SUMMARY:
The purpose of this study is to determine whether strength training can be used as a viable exercise modality for the purpose of inducing fat loss.

DETAILED DESCRIPTION:
Aerobic exercise (AE) is commonly recommended as the most effective exercise modality for weight loss. The Centers for Disease Control (CDC) recommends 150 minutes of AE for weight maintenance, and an unspecified greater amount required for weight loss. Similarly, the American College of Sports Medicine (ACSM) position stand on physical activity for weight loss recommends 150-250 minutes per week of moderate intensity physical activity. While the ACSM promotes resistance training (RT) as a means of increasing fat free mass, which should lead to improved body composition, it does not promote RT for losing significant amounts of body fat. Similarly, the CDC physical activity guidelines for weight loss do not mention RT at all as a viable exercise modality for weight loss. This is not surprising, as there is a paucity of research examining the effects of RT on weight loss. Furthermore, the few studies that have explored RT for weight loss generally show that it is ineffective. The effectiveness of any weight loss program is dependent on the size of the caloric deficit that is created over time, and since AE generally burns more calories per unit of time than RT, it stands to reason that AE would be the most commonly prescribed type of exercise for weight loss. Contributing to the exclusion of RT for weight loss is a widespread belief among dietitians, nutritionists and exercise professionals that it is not possible to induce muscle growth while in a caloric deficit, and since the creation of a caloric deficit is essential for fat loss, the use of RT for muscle growth in a caloric deficit is counter intuitive.

However, RT has been shown to elevate resting metabolism for an extended period of time following cessation of the training session. Additionally, having a greater muscle mass should lead to a greater resting metabolism. Unlike RT, chronic AE performed in a caloric deficit (which is often the recommendation for effective weight loss) has the potential to lead to significant decreases in muscle mass, thereby hampering improvements in body composition. Ideally, a program designed to improve body composition should do so through fat losses alone, with muscle mass being maintained or increased.

Several reasons could exist for the lack of effectiveness of RT shown in most studies. These reasons include, but are not limited to, 1) Body mass being the measured outcome and not body composition, 2) lack of control and/or measurement of caloric intake, 3) failure to adjust dietary protein needs to support muscle growth, 4) ineffective RT program design. Case studies of clients from our lab have routinely shown that profound decreases in bodyfat can be induced with RT as the exclusive form of exercise. Furthermore, these decreases in bodyfat occur with concomitant increases in muscle mass, while in a caloric deficit. Therefore, the specific aims of this proposal are:

1. To determine whether RT combined with dietary intervention (RT+DIET) results in greater decreases in fat mass than (RT) or dietary intervention (DIET) alone.
2. To determine whether RT combined with dietary intervention (RT+DIET) results in greater improvements in body composition than (RT) or dietary intervention (DIET) alone.
3. To determine whether concomitant increases in muscle mass and decreases in fat mass can occur while in a caloric deficit.

The goal of this project is to serve to generate pilot data to determine whether RT can be used as a viable exercise mode for fat loss and muscle gain. We will then pursue funding for a subsequent study that compares the effects of RT versus AE on body composition and fat loss when 1) the caloric intake is monitored to ensure the creation of a caloric deficit, and 2) dietary protein is appropriately increased to support muscle retention/growth.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-29.9 normally menstruating bodyfat >30%

Exclusion Criteria:

* currently dieting to lose weight currently engaged in structured exercise using dietary weight loss supplements Resting Metabolic Rate not within 10% of predicted value

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Fat Free Mass | 0 and 16 weeks
  Fat Free Mass as measured from DXA and recorded in Kg
Change in Fat Mass | 0, 4, 8, 12, 16 weeks
  Fat Mass as measured from DXA and recorded in Kg
Change in Resting Metabolic Rate | 0 and 16 weeks
  Resting Metabolic Rate measured via indirect calorimetry and recorded in kcal / day
Change in Visceral Fat | 0, 4, 8, 12, 16 weeks
  Fat in the Visceral Depot measured from DXA and recorded in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Miller, PhD, Principal Investigator — George Washington University SPH

IPD SHARING:
Plan to Share IPD: No